CLINICAL TRIAL: NCT06891313
Title: Evaluation of Endosseous Implants in One Stage Ridge Splitting Using the Conventional Technique Versus the Use of Piezo Surgery in the Posterior Mandible Region (Randomized Clinical Trial)
Brief Title: One Stage Ridge Splitting Using 2 Different Techniques in the Posterior Mandible
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohannad Ahmed Ismail, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000-0001-6142-0568
Record Dates: First submitted 2025-02-16; First posted 2025-03-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Ridge Augmentation; Bone Augmentation
Keywords: ridge augmentation; One stage ridge splitting in posterior mandible.; Piezo Surgery
MeSH Terms: interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The patients were randomly allocated into two groups utilizing Random Allocation Software version 2.0. then the allocation was concealed in opaque sealed envelopes. In the study group (A) Piezo Surgery inserts are going to be used to create alveolar bone osteotomies, while in the control group (B) bone discs are going to be used. All procedures were performed by one surgeon in both groups, the allocation was revealed to the operator just before the surgery. On the other hand, the patients, outcome assessor and the statistician who analyzed the collected data and performed the statistical analysis were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group A: Piezo Surgery. (Active Comparator): Piezo surgery bone inserts is used to cut crestal osteotomy in the center of the alveolar bone ridge bucco-lingual traversing the compact bone into the spongiosa Followed by two semi vertical osteotomies at least 1.5mm away from the adjacent teeth.
  Interventions: Device: Piezo Surgery.
- Control Group B: Bone Discs. (Active Comparator): Bone discs diameter 7mm mounted on contra angled 1:1 is used to cut crestal osteotomy in the center of the alveolar bone ridge bucco-lingual traversing the compact bone into the spongiosa, followed by two semi vertical osteotomies at least 1.5mm away from the adjacent teeth using bone discs diameter 6.5mm mounted on external irrigation straight hand piece.
  Interventions: Procedure: Bone Discs

INTERVENTIONS:
Device: Piezo Surgery. — Using bone cutting inserts.
  Arms: Study Group A: Piezo Surgery.
Procedure: Bone Discs — Selected bone discs diameters mounted on contra angled hand piece and external irrigation hand piece at gear ratio 1:1.
  Arms: Control Group B: Bone Discs.

SUMMARY:
The selected patients will be informed of the nature of the research work and informed consent will be obtained.

The control group ridge splitting with simultaneous implants using the conventional technique and study group ridge splitting with simultaneous implants using the piezo surgery.

* Pre operative procedures Patients of both groups will be subjected to CBCT.
* Intra operative procedures (for both groups) followed by CBCT will be taken for every patient after 4 months.
* Infiltration local anesthesia will be given to the patient (Articaine 4% 1:100 000 epinephrine).

Both the study and control group will receive:

* In Recipient site, incision of full thickness mucoperiosteal flap inorder to obtain, three-line pyramidal flap, followed by flap reflection.
* The defective site is reevaluated.
* Flap advancement using periosteal releasing incision.
* In the Study group: Piezo surgery bone inserts are used.
* In the Control group: Bone discs diameter are used.
* Followed by bone chisels.
* The point and pilot implant drills are used followed by the sequential use of bone expanders. Based on the preexisting bone, the defect morphology and bone quality. The implant is submerged below the alveolar crest.
* The fixture is inserted submerged below the alveolar bone crest followed by bone smoothening and roundation under external saline irrigation at recommended speed of 38000rpm and gear ratio 1:1 calibrated on fesiodespenser.
* Xenogenic bone particle size of 0.5 mm to 1mm is going to be condensed into the dead space.
* Recheck adequate flap advancement.
* Double line closure using horizontal mattress sutures followed by interrupted sutures on top to allow contact area and wound edge eversion.

DETAILED DESCRIPTION:
-The selected patients will be informed of the nature of the research work and informed consent will be obtained then randomized in equal proportions between, control group ridge splitting with simultaneous implants using the conventional technique and study group ridge splitting with simultaneous implants using the piezo surgery.

* Pre operative procedures Patients of both groups will be subjected to CBCT (diagnostic for upper arch), Diagnostic wax-up and stent fabrication.
* Intra operative procedures (for both groups) followed by CBCT will be taken for every patient after 4 months.
* Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
* Infiltration local anesthesia will be given to the patient (Articaine 4% 1:100 000 epinephrine).

Both the study and control group will receive:

* In Recipient site, using 15C blade on Bard Parker handle incision of full thickness mucoperiosteal flap inorder to obtain, three-line pyramidal flap, reflection using mucoperiosteal elevator molt 9.
* The defective site is reevaluated after its primary evaluation on CBCT using UNC periodontal probe.
* Flap advancement using periosteal releasing incision inorder to allow later tension free flap closure.
* In the Study group: Piezo surgery bone inserts is used to cut crestal osteotomy in the center of the alveolar bone ridge bucco-lingual traversing the compact bone into the spongiosa Followed by two semi vertical osteotomies at least 1.5mm away from the adjacent teeth.
* In the Control group: Bone discs diameter 7mm mounted on contra angled 1:1 is used to cut crestal osteotomy in the center of the alveolar bone ridge bucco-lingual traversing the compact bone into the spongiosa Followed by two semi vertical osteotomies at least 1.5mm away from the adjacent teeth using bone discs diameter 6.5mm mounted on external irrigation straight hand piece.
* First, the spatula bone chisels are used to make sure of extension of osteotomies into the spongy bone in addition to, adequate free of the cut corners, followed by sequential use of tapered bi-angled bone chisels and hammering with bone mallet 3mm shorter than the length of the proposed implant to gain adequate 1ry stability with concurrent support of the buccal plate of bone as well as the mandible by the assistant.
* The point and pilot implant drills are used followed by the sequential use of bone expanders diameters 2.6, 3, 3.4, 3.8 to place an implant of diameter 3.7 or 4.1mm. Based on the preexisting bone, the defect morphology and bone quality. The implant is submerged about 2mm to 3mm below the alveolar crest to compensate for crestal bone resorption.
* Following partial immobilization of the buccal bone segment either book or island pattern. The fixture is inserted submerged below the alveolar bone crest by 2mm to 3mm. Followed by bone smoothening and roundation using large round diamond stone mounted on straight hand piece with external saline irrigation at recommended speed of 38000rpm and gear ratio 1:1 calibrated on fesiodespenser. To avoid soft tissue irritation.
* Xenogenic bone particle size of 0.5 mm to 1mm is going to be condensed into the dead space. To act as a scaffold for the formation of autogenous bone.
* Recheck adequate flap advancement by visualizing passive flap approximation, to allow tension free closure.
* Double line closure using horizontal mattress placed 5mm away from flap margins followed by interrupted sutures on top to allow contact area which is preferred to point contact and wound edge eversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular residual alveolar bone height not less than 8 mm.
* Alveolar bone width from 5mm to 3mm.
* Both genders.
* At least single missing tooth.
* Previous failed implants.
* Tapered or cylinder cross sectioned alveolar bone defect pattern.

Exclusion Criteria:

* Heavy smokers more than 20 cigarettes per day.
* Patients with bone disease that may affect normal healing, example; hyperparathyroidism.
* Patients had radiotherapy and chemotherapy in head and neck.
* Patients had neoplasms in sites to be grafted.
* Patients with Metabolic diseases uncontrolled diabetic patients, Glycated hemoglobin (Hb A1c) more than 7 mg\dl.
* Pregnant females.
* Patients with Para functional habits, apprehensive and non-cooperative.
* Bone pathology related to the site to be grafted.
* Psychological problems, stress situation (socially or professionally), emotional instability, and unrealistic patients' expectations.
* Intraoral soft and hard tissue pathology.
* Systemic condition that contraindicates implant placement.
* Under the age of 18 years.
* Hourglass defects or defects with bone concavities and or undercuts.

Ages: 20 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Bone Quantity of bone gain. | At 4 months from ridge augmentation.
  Measured using linear measurements from Cone Beam Computed Tomography in millimeters.

SECONDARY OUTCOMES:
Soft tissue dehiscence. | baseline 1st Week.
  Exposure of the augmented site. Written Binary Numerical.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aghaloo TL, Moy PK. Which hard tissue augmentation techniques are the most successful in furnishing bony support for implant placement? Int J Oral Maxillofac Implants. 2007;22 Suppl:49-70. PMID 18437791
- [Background] Jensen OT, Bell W, Cottam J. Osteoperiosteal flaps and local osteotomies for alveolar reconstruction. Oral Maxillofac Surg Clin North Am. 2010 Aug;22(3):331-46, vi. doi: 10.1016/j.coms.2010.04.003. PMID 20713266
- [Background] Bravi F, Bruschi GB, Ferrini F. A 10-year multicenter retrospective clinical study of 1715 implants placed with the edentulous ridge expansion technique. Int J Periodontics Restorative Dent. 2007 Dec;27(6):557-65. PMID 18092450
- [Background] Tolstunov L, Hamrick JFE, Broumand V, Shilo D, Rachmiel A. Bone Augmentation Techniques for Horizontal and Vertical Alveolar Ridge Deficiency in Oral Implantology. Oral Maxillofac Surg Clin North Am. 2019 May;31(2):163-191. doi: 10.1016/j.coms.2019.01.005. PMID 30947846
- [Background] Tolstunov L. Classification of the alveolar ridge width: implant-driven treatment considerations for the horizontally deficient alveolar ridges. J Oral Implantol. 2014 Jul;40 Spec No:365-70. doi: 10.1563/aaid-joi-D-14-00023. Epub 2014 Feb 27. PMID 24575743
- [Background] Hammerle CH, Jung RE. Bone augmentation by means of barrier membranes. Periodontol 2000. 2003;33:36-53. doi: 10.1046/j.0906-6713.2003.03304.x. No abstract available. PMID 12950840
- [Background] Urban IA, Nagursky H, Lozada JL. Horizontal ridge augmentation with a resorbable membrane and particulated autogenous bone with or without anorganic bovine bone-derived mineral: a prospective case series in 22 patients. Int J Oral Maxillofac Implants. 2011 Mar-Apr;26(2):404-14. PMID 21483894
- [Background] Urban IA, Nagursky H, Lozada JL, Nagy K. Horizontal ridge augmentation with a collagen membrane and a combination of particulated autogenous bone and anorganic bovine bone-derived mineral: a prospective case series in 25 patients. Int J Periodontics Restorative Dent. 2013 May-Jun;33(3):299-307. doi: 10.11607/prd.1407. PMID 23593623
- [Background] Pellegrino G, Lizio G, Corinaldesi G, Marchetti C. Titanium Mesh Technique in Rehabilitation of Totally Edentulous Atrophic Maxillae: A Retrospective Case Series. J Periodontol. 2016 May;87(5):519-28. doi: 10.1902/jop.2016.150432. Epub 2016 Jan 12. PMID 26759078
- [Background] Misch CM. Comparison of intraoral donor sites for onlay grafting prior to implant placement. Int J Oral Maxillofac Implants. 1997 Nov-Dec;12(6):767-76. PMID 9425757
- [Background] Montazem A, Valauri DV, St-Hilaire H, Buchbinder D. The mandibular symphysis as a donor site in maxillofacial bone grafting: a quantitative anatomic study. J Oral Maxillofac Surg. 2000 Dec;58(12):1368-71. doi: 10.1053/joms.2000.18268. PMID 11117684
- [Background] Clavero J, Lundgren S. Ramus or chin grafts for maxillary sinus inlay and local onlay augmentation: comparison of donor site morbidity and complications. Clin Implant Dent Relat Res. 2003;5(3):154-60. doi: 10.1111/j.1708-8208.2003.tb00197.x. PMID 14575631
- [Background] Pourabbas R, Nezafati S. Clinical results of localized alveolar ridge augmentation with bone grafts harvested from symphysis in comparison with ramus. J Dent Res Dent Clin Dent Prospects. 2007 Spring;1(1):7-12. doi: 10.5681/joddd.2007.002. Epub 2007 Jun 10. PMID 23277827